CLINICAL TRIAL: NCT00622869
Title: A 24 Month, Multicenter, Open-label, Randomized, Controlled Study to Evaluate the Efficacy and Safety of Concentration-controlled Everolimus to Eliminate or to Reduce Tacrolimus Compared to Tacrolimus in de Novo Liver Transplant Recipients
Brief Title: Efficacy and Safety of Concentration-controlled Everolimus to Eliminate or to Reduce Tacrolimus Compared to Tacrolimus in de Novo Liver Transplant Recipients
Acronym: RAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001H2304; 2007-001821-85 (EudraCT Number)
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Liver Transplantation
Keywords: Liver transplantation; everolimus; calcineurin inhibitors; tacrolimus; renal function; MDRD formula; progression of fibrosis
MeSH Terms: interventions — Tacrolimus; Everolimus; Adrenal Cortex Hormones

ARMS (3):
- Everolimus + reduced tacrolimus (Experimental): Low dose tacrolimus (tacrolimus reduced) + everolimus + corticosteroids.
  Interventions: Drug: Tacrolimus (reduced tacrolimus); Drug: Everolimus (reduced tacrolimus); Drug: Corticosteroids
- Tacrolimus elimination (Experimental): Low-dose tacrolimus (until Month 4, then tacrolimus eliminated) + everolimus + corticosteroids.
  Interventions: Drug: Tacrolimus (tacrolimus elimination); Drug: Everolimus (tacrolimus elimination); Drug: Corticosteroids
- Tacrolimus control (Active Comparator): Control dose tacrolimus + corticosteroids.
  Interventions: Drug: Tacrolimus (tacrolimus control); Drug: Corticosteroids

INTERVENTIONS:
Drug: Tacrolimus (reduced tacrolimus) — After everolimus whole blood trough levels were confirmed to be in the target range of 3-8 ng/mL, tacrolimus tapering began, achieving a target tacrolimus whole blood trough level of 3-5 ng/mL by 3 weeks after randomization, a level which was maintained for the duration of the study.
  Other Names: FK-506; fujimycin; Prograf; Advagraf; Protopic
  Arms: Everolimus + reduced tacrolimus
Drug: Tacrolimus (tacrolimus elimination) — After everolimus whole blood trough levels were confirmed to be in the target range of 3-8 ng/mL, tacrolimus tapering began, achieving a target tacrolimus whole blood trough level of 3-5 ng/mL by 3 weeks after randomization. Tacrolimus elimination was started beginning at Month 4. Tacrolimus was tapered after everolimus whole blood trough levels were within the target range of 6-10 ng/mL. Tacrolimus was completely eliminated by the end of Month 4.
  Other Names: FK-506; fujimycin; Prograf; Advagraf; Protopic
  Arms: Tacrolimus elimination
Drug: Tacrolimus (tacrolimus control) — Tacrolimus trough levels were targeted to be maintained at 8-12 ng/mL until Month 4. At Month 4, tacrolimus whole blood trough levels were decreased to a target trough level of 6-10 ng/mL for the remainder of the study.
  Other Names: FK-506; fujimycin; Prograf; Advagraf; Protopic
  Arms: Tacrolimus control
Drug: Everolimus (reduced tacrolimus) — Everolimus was started within 24 hours of randomization at a dose of 1.0 mg twice a day (bid, 2 mg daily dose). The dose was adjusted to maintain everolimus trough blood levels between 3-8 ng/mL for the duration of the study.
  Other Names: RAD-001; Zortress; Certican; Afinitor
  Arms: Everolimus + reduced tacrolimus
Drug: Everolimus (tacrolimus elimination) — Everolimus was started within 24 hours of randomization at a dose of 1.0 mg twice a day (bid, 2 mg daily dose). The dose was adjusted to maintain everolimus trough blood levels between 3-8 ng/mL until Month 4; beginning with Month 4, the dose was adjusted to maintain everolimus trough blood levels between 6-10 ng/mL.
  Other Names: RAD-001; Zortress; Certican; Afinitor
  Arms: Tacrolimus elimination
Drug: Corticosteroids — For patients in all groups, corticosteroids were initiated at or prior to the time of transplantation according to local practice. Corticosteroids could be used for the duration of the study but could not be eliminated before Month 6.

SUMMARY:
This trial was designed to address important issues that impact recipients of liver allografts as well as clinicians, ie, renal function, reduction or discontinuation of tacrolimus early post-transplantation, and progression rate of fibrosis in hepatitis C virus (HCV) positive patients.

DETAILED DESCRIPTION:
This 24-month study consisted of a screening period, a baseline period (3 to 7 days post-transplantation) followed by a run-in period that ended on the day of randomization at 30 days (± 5 days) post-transplantation. Patients were screened for eligibility prior to liver transplantation. Patients who had undergone successful liver transplantation were initiated on a tacrolimus-based regimen that included corticosteroids and entered the baseline period (between 3 and 7 days post-transplantation). At 30 (± 5) days post-transplantation, patients who met additional randomization inclusion/exclusion criteria were randomized into the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent and adhere to study regimen.
* Recipients who are 18-70 years of age of a primary liver transplant from a deceased donor.
* Recipients who have been initiated on an immunosuppressive regimen that contains corticosteroids and tacrolimus, 3-7 days post-transplantation.
* Confirmed recipient hepatitis C virus (HCV) status at Screening (either by antibody or by PCR (polymerase chain reaction).
* Allograft is functioning at an acceptable level by the time of randomization as defined by protocol specific laboratory values.
* Abbreviated Modification of Diet in Renal Disease estimated glomerular filtration rate (MDRD eGFR) ≥ 30 mL/min/1.73m2. Results obtained within 5 days prior to randomization are acceptable, however, no sooner than Day 25 post-transplantation.
* Verification of at least 1 tacrolimus trough level of ≥ 8 ng/mL in the week prior to randomization. Investigators should make adjustments in tacrolimus dosing to continue to target trough levels above 8 ng/mL prior to randomization.

Exclusion Criteria

* Patients who are recipients of multiple solid organ or islet cell tissue transplants, or have previously received an organ or tissue transplant. Patients who have a combined liver-kidney transplant.
* Recipients of a liver from a living donor, or of a split liver.
* History of malignancy of any organ system within the past 5 years whether or not there is evidence of local recurrence or metastases, other than non-metastatic basal or squamous cell carcinoma of the skin, or HCC (hepatocellular carcinoma) (see next criteria).
* Hepatocellular carcinoma that does not fulfill Milan criteria (1 nodule ≤ 5 cm, 2-3 nodules all < 3 cm) at the time of transplantation as per explant histology of the recipient liver.
* Any use of antibody induction therapy.
* Patients with a known hypersensitivity to the drugs used on study or their class, or to any of the excipients.
* Patients who are recipients of ABO incompatible transplant grafts.
* Recipients of organs from donors who test positive for Hepatitis B surface antigen or HIV are excluded.
* Patients who have any surgical or medical condition, which in the opinion of the investigator, might significantly alter the absorption, distribution, metabolism and excretion of study drug.
* Women of child-bearing potential (WOCBP).
* Patients with any history of coagulopathy or medical condition requiring long-term anticoagulation which would preclude liver biopsy after transplantation. (Low dose aspirin treatment or interruption of chronic anticoagulant is allowed).

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 719 (Actual)
Dates: Start 2008-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (82):
- United States (23):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Newark, New Jersey
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
- Argentina (3):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, San Martín, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
- Australia (4):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Belgium (3):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Brazil (5):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Blumenau, Santa Catarina
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (4):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- Colombia (3):
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Cali
  - Novartis Investigative Site, Medellín
- Novartis Investigative Site, Prague, Czech Republic, Czechia
- France (7):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Villejuif
- Germany (8):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Regensburg
- Novartis Investigative Site, Budapest, Hungary
- Novartis Investigative Site, Dublin, Ireland, Ireland
- Israel (2):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Tel Aviv
- Italy (5):
  - Novartis Investigative Site, Pisa, Italy
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
- Novartis Investigative Site, Rotterdam, Netherlands
- Novartis Investigative Site, Moscow, Russia
- Spain (7):
  - Novartis Investigative Site, Barakaldo, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Majadanonda, Madrid
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Valencia, Valencia
- Novartis Investigative Site, Stockholm, Sweden
- United Kingdom (2):
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, London

REFERENCES:
- [Derived] Charlton M, Rinella M, Patel D, McCague K, Heimbach J, Watt K. Everolimus Is Associated With Less Weight Gain Than Tacrolimus 2 Years After Liver Transplantation: Results of a Randomized Multicenter Study. Transplantation. 2017 Dec;101(12):2873-2882. doi: 10.1097/TP.0000000000001913. PMID 28817434
- [Derived] Fischer L, Saliba F, Kaiser GM, De Carlis L, Metselaar HJ, De Simone P, Duvoux C, Nevens F, Fung JJ, Dong G, Rauer B, Junge G; H2304 Study Group. Three-year Outcomes in De Novo Liver Transplant Patients Receiving Everolimus With Reduced Tacrolimus: Follow-Up Results From a Randomized, Multicenter Study. Transplantation. 2015 Jul;99(7):1455-62. doi: 10.1097/TP.0000000000000555. PMID 26151607
- [Derived] Saliba F, De Simone P, Nevens F, De Carlis L, Metselaar HJ, Beckebaum S, Jonas S, Sudan D, Fischer L, Duvoux C, Chavin KD, Koneru B, Huang MA, Chapman WC, Foltys D, Dong G, Lopez PM, Fung J, Junge G; H2304 Study Group. Renal function at two years in liver transplant patients receiving everolimus: results of a randomized, multicenter study. Am J Transplant. 2013 Jul;13(7):1734-45. doi: 10.1111/ajt.12280. Epub 2013 May 28. PMID 23714399

RESULTS

PARTICIPANT FLOW:
Groups:
- Tacrolimus Control Arm: Control dose tacrolimus + corticosteroids.
Period: Overall Study
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination | Tacrolimus Control Arm
Started | 245 | 231 | 243
Completed | 202 | 174 | 204
Not Completed | 43 | 57 | 39
Not completed — Subject Withdrew Consent | 13 | 17 | 11
Not completed — Administrative Problems | 11 | 17 | 13
Not completed — Death | 12 | 15 | 10
Not completed — Lost to Follow-up | 2 | 4 | 2
Not completed — Graft Loss | 5 | 3 | 2
Not completed — Missing | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination | Tacrolimus Control Arm | Total
Number analyzed (Participants) | 245 | 231 | 243 | 719
Age Continuous [Mean (Standard Deviation); unit: years] | 53.6 (9.2) | 53.2 (10.8) | 54.5 (8.7) | 53.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 67 | 64 | 196
  Male | 180 | 164 | 179 | 523

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Composite Efficacy Failure From Randomization to Month 12
Description: Composite efficacy failure was defined as treated biopsy proven acute rejection (tBPAR), graft loss, or death. A BPAR was defined as an acute rejection confirmed by biopsy with a Rejection Activity Index (RAI) score ≥ 3. tBPAR was defined as a BPAR which was treated with anti-rejection therapy. The RAI is used to score liver biopsies with acute rejection and is composed of 3 categories (portal inflammation, bile duct inflammation damage, venous endothelial inflammation) each scored on a scale of 0 (absent) to 3 (severe) by a trained pathologist. The total RAI score = the sum of the scores of the 3 categories and ranges from 0 to 9, with a higher score indicating greater rejection. The graft was presumed to be lost on the day the patient was newly listed for a liver graft, they received a graft re-transplant, or they died.
  The incidence rates of composite efficacy failure were estimated with a Kaplan-Meier product-limit formula.
Time Frame: Randomization to Month 12
Population: Intent-to-treat population: All randomized patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination | Tacrolimus Control Arm
Number analyzed (Participants) | 245 | 231 | 243
Percentage of participants | 6.7 | 24.2 | 9.7

2. Secondary Outcome: Incidence Rate of Composite Efficacy Failure From Randomization to Month 24
Description: Composite efficacy failure was defined as treated biopsy proven acute rejection (tBPAR), graft loss, or death.
  The incidence rates of composite efficacy failure were estimated with a Kaplan-Meier product-limit formula.
Time Frame: Randomization to Month 24
Population: Intent-to-treat population: All randomized patients.
Measure: Number; unit: Percentage
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination | Tacrolimus Control Arm
Number analyzed (Participants) | 245 | 231 | 243
Percentage | 10.3 | 26.0 | 12.5

3. Secondary Outcome: Incidence Rate of Treated Biopsy Proven Acute Rejection (tBPAR) at Months 12 and 24
Description: tBPAR was defined as an acute rejection confirmed by biopsy with a Rejection Activity Index (RAI) score ≥ 3, which was treated with anti-rejection therapy. Liver biopsies were collected for all cases of suspected acute rejection preferably within 24 hours, at the latest within 48 hours, whenever clinically possible. The RAI is used to score liver biopsies with acute rejection and is composed of 3 categories (portal inflammation, bile duct inflammation damage, venous endothelial inflammation) each scored on a scale of 0 (absent) to 3 (severe) by a trained pathologist. The total RAI score = the sum of the scores of the 3 categories and ranges from 0 to 9, with a higher score indicating greater rejection. The graft was presumed to be lost on the day the patient was newly listed for a liver graft, they received a graft re-transplant, or they died.
  The incidence rates of tBPAR were estimated with a Kaplan-Meier product-limit formula.
Time Frame: Randomization to Month 24
Population: Intent-to-treat population: All randomized patients.
Measure: Number; unit: Percentage
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination | Tacrolimus Control Arm
Number analyzed (Participants) | 245 | 231 | 243
Percentage
  Month 12 | 3.0 | 18.8 | 7.2
  Month 24 | 4.8 | 19.9 | 7.7

4. Secondary Outcome: Change in Renal Function From Randomization to Months 12 and 24
Description: Change in renal function was assessed by the estimated Glomerular Filtration Rate (eGFR) using the abbreviated (4 variables) Modification of Diet in Renal Disease (MDRD-4) formula which was developed by the MDRD Study Group and has been validated in patients with chronic kidney disease. The MDRD-4 formula used for the eGFR calculation is: eGFR (mL/min/1.73m^2) = 186.3*(C^-1.154)*(A^-0.203)*G*R, where C is the serum concentration of creatinine (mg/dL), A is age (years), G=0.742 when gender is female, otherwise G=1, R=1.21 when race is black, otherwise R=1.
  The changes in renal function were analyzed via analysis of covariance (ANCOVA) with treatment, pre-transplant hepatitis C virus status and randomization eGFR as covariates. Based on these ANCOVA analyses, the least-squares mean and standard errors of change were reported.
Time Frame: Randomization to Month 24
Population: Intent-to-treat population: All randomized patients.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination | Tacrolimus Control Arm
Number analyzed (Participants) | 245 | 231 | 243
mL/min/1.73m^2
  Month 12 (N=244, 231, 243) | -2.23 (1.54) | -1.51 (1.58) | -10.73 (1.54)
  Month 24 (N=245, 231, 243) | -7.94 (1.53) | -4.19 (1.58) | -14.60 (1.54)

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were followed until resolution or judged permanent. Serious AEs occurring after transplantation, until 30 days after study medication (SM) discontinuation, or > 4 weeks after study discontinuation if related to SM were reported.
Description: Safety population: All patients who received at least 1 dose of randomized study medication.
  Adverse events up to Month 24 were reported.
Groups:
- Tacrolimus Elimination: Low dose tacrolimus (until Month 4, then tacrolimus eliminated) + everolimus + corticosteroids
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination | Tacrolimus Control Arm
Serious Adverse Events (participants affected / at risk) | 138/245 | 152/229 | 131/242
Other Adverse Events (participants affected / at risk) | 218/245 | 194/229 | 205/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Reduced Tacrolimus (N=245) | Tacrolimus Elimination (N=229) | Tacrolimus Control Arm (N=242)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 5
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 6 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 2
Angina pectoris (Cardiac disorders) | 2 | 0 | 3
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 3 | 0 | 3
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0
Hepato-lenticular degeneration (Congenital, familial and genetic disorders) | 0 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 2 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 5 | 11 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 7 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 4 | 3 | 2
Colitis (Gastrointestinal disorders) | 0 | 3 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 11 | 4
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 0 | 1
Femoral hernia (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Gingival erosion (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Hernial eventration (Gastrointestinal disorders) | 2 | 2 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 1 | 3
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 2 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 2 | 2 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatic mass (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Spigelian hernia (Gastrointestinal disorders) | 0 | 1 | 1
Tongue oedema (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 3 | 3 | 2
Umbilical hernia, obstructive (Gastrointestinal disorders) | 2 | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 6 | 0
Asthenia (General disorders) | 1 | 3 | 0
Device dislocation (General disorders) | 0 | 1 | 1
Device occlusion (General disorders) | 1 | 0 | 0
Drug ineffective (General disorders) | 0 | 1 | 0
Feeling jittery (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 1
Hernia obstructive (General disorders) | 0 | 1 | 0
Impaired healing (General disorders) | 1 | 1 | 0
Malaise (General disorders) | 1 | 1 | 1
Medical device complication (General disorders) | 1 | 0 | 1
Multi-organ failure (General disorders) | 5 | 1 | 4
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 14 | 20 | 7
Sensation of foreign body (General disorders) | 1 | 0 | 0
Spinal pain (General disorders) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 3 | 7 | 6
Bile duct stone (Hepatobiliary disorders) | 1 | 3 | 1
Biliary cast syndrome (Hepatobiliary disorders) | 0 | 0 | 2
Biliary cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Biliary cirrhosis primary (Hepatobiliary disorders) | 1 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1 | 0
Biliary ischaemia (Hepatobiliary disorders) | 2 | 2 | 3
Biliary tract disorder (Hepatobiliary disorders) | 0 | 0 | 1
Biloma (Hepatobiliary disorders) | 3 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 11 | 11 | 6
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Cholangitis chronic (Hepatobiliary disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 1
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 6 | 3 | 5
Chronic hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic artery stenosis (Hepatobiliary disorders) | 0 | 4 | 2
Hepatic artery thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic necrosis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic vein occlusion (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 2 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 1 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 2 | 2 | 1
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 2 | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 1 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 2
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Liver transplant rejection (Immune system disorders) | 4 | 24 | 9
Overlap syndrome (Immune system disorders) | 0 | 0 | 1
Serum sickness (Immune system disorders) | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0
Abscess intestinal (Infections and infestations) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 1
Biliary sepsis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 2
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 4 | 0 | 3
Cholangitis suppurative (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 3 | 2 | 1
Device related infection (Infections and infestations) | 0 | 1 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Enterobacter sepsis (Infections and infestations) | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 1
Enterococcal sepsis (Infections and infestations) | 1 | 1 | 2
Erysipelas (Infections and infestations) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 2 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 5 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 3 | 0 | 0
H1N1 influenza (Infections and infestations) | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 10 | 7 | 7
Herpes virus infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 1
Herpes zoster oticus (Infections and infestations) | 0 | 1 | 0
Histoplasmosis (Infections and infestations) | 0 | 1 | 0
Incision site infection (Infections and infestations) | 0 | 1 | 0
Infected bites (Infections and infestations) | 1 | 0 | 0
Infected cyst (Infections and infestations) | 1 | 2 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Infectious peritonitis (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1
Klebsiella infection (Infections and infestations) | 1 | 1 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1
Liver abscess (Infections and infestations) | 1 | 1 | 2
Localised infection (Infections and infestations) | 1 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 3 | 1
Meningitis cryptococcal (Infections and infestations) | 1 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0
Peritoneal abscess (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 9 | 4
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1
Pneumonia herpes viral (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 2
Pyelonephritis (Infections and infestations) | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 2
Septic shock (Infections and infestations) | 3 | 3 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Sinusitis aspergillus (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Splenic abscess (Infections and infestations) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 3 | 2
Urosepsis (Infections and infestations) | 0 | 1 | 0
Wound abscess (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 2 | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 3 | 3 | 6
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Chemical peritonitis (Injury, poisoning and procedural complications) | 2 | 2 | 1
Complications of transplanted heart (Injury, poisoning and procedural complications) | 0 | 0 | 1
Complications of transplanted liver (Injury, poisoning and procedural complications) | 1 | 4 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0
Graft dysfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Graft loss (Injury, poisoning and procedural complications) | 1 | 2 | 2
Hepatic haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Hypoinsulinaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 9 | 7 | 5
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 0 | 0
Liver graft loss (Injury, poisoning and procedural complications) | 2 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 2 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 2 | 2 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 2 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood lactic acid increased (Investigations) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 0
Chest X-ray abnormal (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 4 | 4 | 5
Immunosuppressant drug level increased (Investigations) | 1 | 1 | 0
Liver function test abnormal (Investigations) | 3 | 4 | 2
Platelet count decreased (Investigations) | 0 | 1 | 0
Renal function test abnormal (Investigations) | 0 | 1 | 1
Transaminases increased (Investigations) | 4 | 1 | 3
Urine output decreased (Investigations) | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2 | 2
Diabetes mellitus malnutrition-related (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 1
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Aphasia (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Cluster headache (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 1 | 1
Critical illness polyneuropathy (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 3 | 0 | 3
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Monoparesis (Nervous system disorders) | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 0
Radiculitis brachial (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 2 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Adjustment disorder (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1
Alcoholism (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 2 | 2 | 0
Drug abuse (Psychiatric disorders) | 1 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 2
Nervousness (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 2
Nephropathy toxic (Renal and urinary disorders) | 1 | 1 | 1
Nephrosclerosis (Renal and urinary disorders) | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 9 | 4 | 7
Renal failure acute (Renal and urinary disorders) | 11 | 3 | 5
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 3 | 0
Ureteric fistula (Renal and urinary disorders) | 0 | 1 | 0
Endometrial dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cholestatic pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Scar (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Colostomy closure (Surgical and medical procedures) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Hyperaemia (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 3
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0
Lymphocele (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Reduced Tacrolimus (N=245) | Tacrolimus Elimination (N=229) | Tacrolimus Control Arm (N=242)
Anaemia (Blood and lymphatic system disorders) | 22 | 26 | 20
Leukopenia (Blood and lymphatic system disorders) | 31 | 23 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 17 | 5
Abdominal pain (Gastrointestinal disorders) | 35 | 29 | 28
Abdominal pain upper (Gastrointestinal disorders) | 13 | 10 | 16
Constipation (Gastrointestinal disorders) | 18 | 16 | 20
Diarrhoea (Gastrointestinal disorders) | 56 | 55 | 58
Nausea (Gastrointestinal disorders) | 36 | 23 | 33
Vomiting (Gastrointestinal disorders) | 20 | 17 | 21
Fatigue (General disorders) | 27 | 22 | 28
Oedema peripheral (General disorders) | 49 | 43 | 31
Pyrexia (General disorders) | 37 | 39 | 23
Cholestasis (Hepatobiliary disorders) | 15 | 7 | 7
Hepatitis C (Infections and infestations) | 25 | 17 | 21
Nasopharyngitis (Infections and infestations) | 24 | 24 | 26
Urinary tract infection (Infections and infestations) | 21 | 16 | 11
Incisional hernia (Injury, poisoning and procedural complications) | 19 | 9 | 15
Blood creatinine increased (Investigations) | 5 | 6 | 18
Hepatic enzyme increased (Investigations) | 13 | 19 | 14
Liver function test abnormal (Investigations) | 16 | 25 | 23
Transaminases increased (Investigations) | 14 | 9 | 9
Decreased appetite (Metabolism and nutrition disorders) | 16 | 6 | 16
Diabetes mellitus (Metabolism and nutrition disorders) | 17 | 8 | 12
Hypercholesterolaemia (Metabolism and nutrition disorders) | 27 | 21 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 12 | 8 | 24
Hyperlipidaemia (Metabolism and nutrition disorders) | 21 | 24 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 20 | 9 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 9 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 19 | 6 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 12 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 13 | 29
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 9 | 23
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 14 | 16
Headache (Nervous system disorders) | 51 | 40 | 53
Tremor (Nervous system disorders) | 23 | 17 | 36
Depression (Psychiatric disorders) | 16 | 9 | 14
Insomnia (Psychiatric disorders) | 16 | 18 | 24
Renal failure (Renal and urinary disorders) | 18 | 12 | 22
Renal impairment (Renal and urinary disorders) | 8 | 7 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 14 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 5 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 6 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13 | 6 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 11 | 6
Pruritus generalised (Skin and subcutaneous tissue disorders) | 13 | 14 | 17
Hypertension (Vascular disorders) | 51 | 35 | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.